CLINICAL TRIAL: NCT02713074
Title: A Comparison Between Povidone-iodine and Normal Saline in Vaginal Cleansing Before Office Hysterosocpy: a Randomized Controlled Trial
Brief Title: Povidone-iodine Versus Saline in Vaginal Cleansing Before Office Hysteroscopy
Acronym: PISOH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI-S
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Postoperative Infection
MeSH Terms: interventions — Povidone-Iodine; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): povidone-iodine group
  Interventions: Drug: povidone-iodine
- Group B (Active Comparator): Normal saline group
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: povidone-iodine — The patients will be subjected to povidone-iodine (Betadine7.5%) for vaginal cleaning before office hysteroscopy
  Arms: Group A
Drug: normal saline — The patients will be subjected to normal saline (Sod. Chloride 0.9%, Nile) for vaginal cleaning
  Arms: Group B

SUMMARY:
The normal saline is used in medicine as an intravenous isotonic infusion and for cleaning wounds. It is a mild but effective cleaning agent and will not harm normal tissue, unlike many stronger antiseptics. It is available and inexpensive in comparison to povidone iodine.

ELIGIBILITY:
Inclusion Criteria:

1 - All women who will subject to office Hysterosocpy for gynecological problems

Exclusion Criteria:

1. All patients have current vaginitis or urinary tract infection before the hysteroscopy
2. Diabetic women.
3. Women with body mass index > 25 kg/m2.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
rate of postoperative vaginal irritation symptoms | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No